CLINICAL TRIAL: NCT02947022
Title: Investigator Initiated Investigational New Drug Application to Study the Effects of IV-Administered Ca-DTPA and Zn-DTPA To Treat Patients With Gadolinium Deposition Disease
Brief Title: Effects of IV-Administered Ca-DTPA and Zn-DTPA To Treat Patients With Gadolinium Deposition Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI left institution.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Hameln Pharma GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-1080
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-02

CONDITIONS: Headache; Cognitive Disturbance; Skin Hyperpigmentation; Arthralgia
Keywords: gadolinium; deposition; GBCA; Extremity Pain; Skin Pain; Chest Wall Pain
MeSH Terms: conditions — Headache; Cognition Disorders; Hyperpigmentation; Arthralgia | interventions — Pentetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Calcium DTPA followed by Zinc DTPA (Experimental): Subjects will receive IV administration of Ca-DTPA on Day 1 and Zn-DTPA on Day 2 at each of treatment time-points. Three identical treatment time-points are scheduled on Month 1, Month 2 and Month 3.
  Interventions: Drug: Calcium DTPA; Drug: Zinc DTPA

INTERVENTIONS:
Drug: Calcium DTPA — On Day 1, 2.5 mL of Ca-DTPA (1 g/5 mL) will be administered over a period of 1 minute. A solution of normal saline will then be administered at a rate of 300 mL/hr over 30 minutes. Patients will be seated with hands lowered to their sides to allow the chelator to dwell slightly in the soft tissues of the hands and feet. Patients will then be moved to a supine position and the infusion rate increased to 750 mL/hr over the next 60 minutes. At 90 minutes the remaining 2.5 mL of Ca-DTPA will administered IV over a period of 1 minute, and the normal saline will continue for the remaining 9 minutes. The IV line will then be removed. Patients will be instructed to drink plenty of fluids that evening.
  The same treatment therapy will consist of 3 time-points, approximately 1 month apart.
  Other Names: Pentetate calcium trisodium injection
Drug: Zinc DTPA — On Day 2, 2.5 mL of Zn-DTPA (1 g/5 mL) will be administered over a period of 1 minute. A solution of normal saline will then be administered at a rate of 300 mL/hr over 30 minutes. Patients will be seated with hands lowered to their sides to allow the chelator to dwell slightly in the soft tissues of the hands and feet. Patients will then be moved to a supine position and the infusion rate increased to 750 mL/hr over the next 60 minutes. At 90 minutes the remaining 2.5 mL of Zn-DTPA will administered IV over a period of 1 minute, and the normal saline will continue for the remaining 9 minutes. The IV line will then be removed. Patients will be instructed to drink plenty of fluids that evening.
  The same treatment therapy will consist of 3 time-points, approximately 1 month apart.
  Other Names: Pentetate zinc trisodium injection

SUMMARY:
Purpose: There are two goals we have for this prospective single arm study; to see an increase in the amount of gadolinium in 24 hour urine collection following each infusion treatment with Calcium and Zinc DTPA, and to see a reduction or elimination of gadolinium deposition disease (GDD) symptoms.

Participants: Twenty (20) patients who are suffering from gadolinium deposition disease (GDD)

Procedures: Over a series of three (3) treatment time-points patients will be treated with IV Ca-DTPA on day one, and Zn-DTPA on day two.

ELIGIBILITY:
Inclusion Criteria: Exhibiting 3 or greater of the following symptoms which must be present after having been administered a GBCA:

* Cognitive disturbance
* Extremity pain
* Headache
* Chest wall pain
* Skin induration
* Skin hyperpigmentation
* Skin pain
* Arthralgia

Exclusion Criteria:

* Pregnant or lactating
* Less than 18 years old
* No evidence of gadolinium (has to have shown previous demonstration of Gd by urine analysis or bone biopsy)
* Known connective tissue disease such as Systemic Lupus Erythematosus or Scleroderma
* Severe hemochromatosis or Wilson's disease
* Glomerular Filtration Rate (GFR) ≤ 60
* Have had an investigational drug within last 30 days
* Unable to give written consent
* Multiple Sclerosis
* Chronic heart failure
* Cirrhosis of the liver

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-10; Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Semelka, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospitals, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Calcium DTPA Followed by Zinc DTPA: Subjects will receive IV administration of Ca-DTPA on Day 1 and Zn-DTPA on Day 2 at each of treatment time-points. Three identical treatment time-points are scheduled on Month 1, Month 2 and Month 3.
  Calcium DTPA: On Day 1, 2.5 mL of Ca-DTPA (1 g/5 mL) will be administered over a period of 1 minute. A solution of normal saline will then be administered at a rate of 300 mL/hr over 30 minutes. Patients will be seated with hands lowered to their sides to allow the chelator to dwell slightly in the soft tissues of the hands and feet. Patients will then be moved to a supine position and the infusion rate increased to 750 mL/hr over the next 60 minutes. At 90 minutes the remaining 2.5 mL of Ca-DTPA will administered IV over a period of 1 minute, and the normal saline will continue for the remaining 9 minutes. The IV line will then be removed. Patients will be instructed to drink plenty of fluids that evening.
  The same treatment therapy will consist of 3 time-points, approximately 1 m
Period: Overall Study
Arm/Group | Calcium DTPA Followed by Zinc DTPA
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study Stopped | 1

BASELINE CHARACTERISTICS:
Population: One patient was enrolled and treated in the trial. The patient did not have any adequate follow up data for analyses.
Arm/Group | Calcium DTPA Followed by Zinc DTPA
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 1 in Gd Level From 24-hour Urine Samples Following Calcium DTPA Administration.
Time Frame: Baseline, Month 1
Population: Data were not analyzed because this study was stopped prematurely.
Groups:
- Calcium DTPA Followed by Zinc DTPA: Subjects will receive IV administration of Ca-DTPA on Day 1 and Zn-DTPA on Day 2 at each of treatment time-points. Three identical treatment time-points are scheduled on Month 1, Month 2 and Month 3.
  Calcium DTPA: On Day 1, 2.5 mL of Ca-DTPA (1 g/5 mL) will be administered over a period of 1 minute. A solution of normal saline will then be administered at a rate of 300 mL/hr over 30 minutes. Patients will be seated with hands lowered to their sides to allow the chelator to dwell slightly in the soft tissues of the hands and feet. Patients will then be moved to a supine position and the infusion rate increased to 750 mL/hr over the next 60 minutes. At 90 minutes the remaining 2.5 mL of Ca-DTPA will administered IV over a period of 1 minute, and the normal saline will continue for the remaining 9 minutes. The IV line will then be removed. Patients will be instructed to drink plenty of fluids that evening.
  The same treatment therapy will consist of 3 time-points, approximately 1 mo
Arm/Group | Calcium DTPA Followed by Zinc DTPA
Number analyzed (Participants) | 0

2. Primary Outcome: Change From Baseline to Month 1 in Gd Level From 24-hour Urine Samples Following Zinc DTPA Administration.
Time Frame: Baseline, Month 1
Population: Data were not analyzed because this study was stopped prematurely.
Arm/Group | Calcium DTPA Followed by Zinc DTPA
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline to Month 2 in Gd Level From 24-hour Urine Samples Following Calcium DTPA Administration.
Time Frame: Baseline, Month 2
Population: Data were not analyzed because this study was stopped prematurely.
Arm/Group | Calcium DTPA Followed by Zinc DTPA
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline to Month 2 in Gd Level From 24-hour Urine Samples Following Zinc DTPA Administration.
Time Frame: Baseline, Month 2
Population: Data were not analyzed because this study was stopped prematurely.
Groups:
- Calcium DTPA Followed by Zinc DTPA: Subjects will receive IV administration of Ca-DTPA on Day 1 and Zn-DTPA on Day 2 at each of treatment time-points. Three identical treatment time-points are scheduled on Month 1, Month 2 and Month 3.
  Calcium DTPA: On Day 1, 2.5 mL of Ca-DTPA (1 g/5 mL) will be administered over a period of 1 minute. A solution of normal saline will then be administered at a rate of 300 mL/hr over 30 minutes. Patients will be seated with hands lowered to their sides to allow the chelator to dwell slightly in the soft tissues of the hands and feet. Patients will then be moved to a supine position and the infusion rate increased to 750 mL/hr over the next 60 minutes. At 90 minutes the remaining 2.5 mL of Ca-DTPA will administered IV over a period of 1 minute, and the normal saline will continue for the remaining 9 minutes. The IV line will then be removed. Patients will be instructed to drink plenty of fluids that evening.
  The same treatment therapy will consist of 3 time-points, approximately 1
Arm/Group | Calcium DTPA Followed by Zinc DTPA
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline to Month 3 in Gd Level From 24-hour Urine Samples Following Calcium DTPA Administration.
Time Frame: Baseline, Month 3
Population: Data were not analyzed because this study was stopped prematurely.
Arm/Group | Calcium DTPA Followed by Zinc DTPA
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline to Month 3 in Gd Level From 24-hour Urine Samples Following Zinc DTPA Administration.
Time Frame: Baseline, Month 3
Population: Data were not analyzed because this study was stopped prematurely.
Arm/Group | Calcium DTPA Followed by Zinc DTPA
Number analyzed (Participants) | 0

7. Secondary Outcome: Change From Baseline to Month 1 in the Pain Score
Description: Patient self-reported pain scores assessed using a Visual Analog Scale (VAS) ranging from 0 to 10 where 0 indicates "no pain", 4 through 6 reflect "moderate pain", and 10 reflects "worst possible pain".
Time Frame: Baseline, Month 1 (Day 7)
Population: Data were not analyzed because this study was stopped prematurely.
Arm/Group | Calcium DTPA Followed by Zinc DTPA
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline to Month 2 in the Pain Score
Description: Patient self-reported pain scores assessed using a VAS ranging from 0 to 10 where 0 indicates "no pain", 4 through 6 reflect "moderate pain", and 10 reflects "worst possible pain".
Time Frame: Baseline, Month 2 (Day 7)
Population: Data were not analyzed because this study was stopped prematurely.
Arm/Group | Calcium DTPA Followed by Zinc DTPA
Number analyzed (Participants) | 0

9. Secondary Outcome: Change From Baseline to Month 3 in the Pain Score
Description: as for outcome 8
Time Frame: Baseline, Month 3 (Day 7)
Population: Data were not analyzed because this study was stopped prematurely.
Arm/Group | Calcium DTPA Followed by Zinc DTPA
Number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline to Month 6 in the Pain Score
Description: as for outcome 8
Time Frame: Baseline, Month 6
Population: Data were not analyzed because this study was stopped prematurely.
Arm/Group | Calcium DTPA Followed by Zinc DTPA
Number analyzed (Participants) | 0

11. Secondary Outcome: Change From Baseline to Month 12 in the Pain Score
Description: as for outcome 8
Time Frame: Baseline, Month 12
Population: Data were not analyzed because this study was stopped prematurely.
Arm/Group | Calcium DTPA Followed by Zinc DTPA
Number analyzed (Participants) | 0

12. Secondary Outcome: Change in American Chronic Pain Association (ACPA) Quality of Life (QOL) Score From Baseline to Month 1
Description: The ACPA QOL is a self-administered questionnaire measuring functionality for people with pain which looks at the ability to function, rather than pain alone and is intended to measure activity levels. The ACPA QOL consists of 10 possibilities ranging from 0 to 10 where 0 represents "Non-functioning" and 10 represents "Normal Quality of Life".
Time Frame: Baseline, Month 1 (day 7)
Population: Data were not analyzed because this study was stopped prematurely.
Arm/Group | Calcium DTPA Followed by Zinc DTPA
Number analyzed (Participants) | 0

13. Secondary Outcome: Change in ACPA QOL Score From Baseline to Month 2
Description: as for outcome 12
Time Frame: Baseline, Month 2 (day 7)
Population: Data were not analyzed because this study was stopped prematurely.
Arm/Group | Calcium DTPA Followed by Zinc DTPA
Number analyzed (Participants) | 0

14. Secondary Outcome: Change in ACPA QOL Score at Month 3
Description: as for outcome 12
Time Frame: Baseline, Month 3 (day 7)
Population: Data were not analyzed because this study was stopped prematurely.
Arm/Group | Calcium DTPA Followed by Zinc DTPA
Number analyzed (Participants) | 0

15. Secondary Outcome: Change in ACPA QOL Score at Month 6
Description: as for outcome 12
Time Frame: Baseline, Month 6
Population: Data were not analyzed because this study was stopped prematurely.
Arm/Group | Calcium DTPA Followed by Zinc DTPA
Number analyzed (Participants) | 0

16. Secondary Outcome: Change in ACPA QOL Score at Month 12
Description: as for outcome 12
Time Frame: Baseline, Month 12
Population: Data were not analyzed because this study was stopped prematurely.
Arm/Group | Calcium DTPA Followed by Zinc DTPA
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Throughout treatment and for 12 days after the last dose (or cessation), an average of 2 weeks.
Arm/Group | Calcium DTPA Followed by Zinc DTPA
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The study was stopped on 1/31/16. Only 1 patient received 1 treatment prior to the study stopping.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT02947022/Prot_SAP_000.pdf